CLINICAL TRIAL: NCT05651438
Title: Investigation of Factors Associated With Pain, Fatigue and Sleep Quality in E-Athletes
Brief Title: Pain, Fatigue and Sleep Quality of E-Athletes
Status: Completed | Type: Observational
Sponsor: Bandırma Onyedi Eylül University (Other)
Responsible Party: Principal Investigator, Melike Sumeyye Ozen, Research Assistant, Bandırma Onyedi Eylül University
Other Study IDs: 2022-84
Record Dates: First submitted 2022-12-05; First posted 2022-12-15 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: E-Athletes
Keywords: E-Athletes; pain; fatigue; sleep quality
MeSH Terms: conditions — Pain; Fatigue; Sleep Initiation and Maintenance Disorders | interventions — Restraint, Physical

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- E-Athletes: E-Athletes who are over the age of 18, have participated in professional matches for at least one year, and have an E-sports license were evaluated.
  Interventions: Other: Assessment

INTERVENTIONS:
Other: Assessment — Assessment of pain, fatigue, sleep quality, physical activity status, and e-sports-specific features

SUMMARY:
E-Sports, which attract great attention in the media and social networks, brings health problems and some risks, depending on the attractiveness of games and the time spent in the digital world. When the investigators examine the literature, although different studies are showing that E-Athletes experience pain and sleep problems, no study examines the factors related to pain and sleep quality together. Therefore, our study was planned to examine the factors associated with pain, fatigue, and sleep quality in E-Athletes.

ELIGIBILITY:
The inclusion criteria were: (1) being between 18 and 35 years of age, (2) being under contract with a professional gaming corporation, (3) being primarily engaged in esports through a computer-based game, (4) having at least one year of professional gaming experience, and (5) volunteering to participate in the study.

The exclusion criteria were: (1) being retired from esports and (2) having any systemic, orthopedic, or neurological disease.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: E-sports players over the age of 18 who have participated in professional matches for at least one year will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Pain assessment | baseline
  The area where the pain is experienced, the situation of applying to a health institution for pain, the situation of applying to a physiotherapist for pain, and pain severity (with the Numerical Rating Scale (NRS) will be questioned. NRS: The number 0 is defined as "no pain" and the number 10 as "unbearable pain".
Fatigue severity | baseline
  Fatigue severity will be evaluated using the Numerical Rating Scale (NRS), where 0 will indicate "no fatigue" and 10 will indicate "worst possible fatigue." Participants will report the degree of fatigue they will have felt during the past 24 hours, reflecting their overall daily experience.
Pittsburgh Sleep Quality Index | baseline
  It is used to assess sleep quality. The total score ranges from 0 to 21. The sleep quality of people with a total score of less than 5 is "good"; For those with more than 5, it means "poor" sleep quality.
Epworth Sleepiness Scale | baseline
  It is used to evaluate daytime sleepiness. The scoring method is the same for all questions, 0 if there is no probability of falling asleep, 1 if there is a low probability of falling asleep, 2 if there is a medium probability, and 3 if there is a high probability of falling asleep. A score of 10 or more indicates the presence of excessive daytime sleepiness.

SECONDARY OUTCOMES:
Demographic variables | baseline
  Age, gender
Esports-related characteristics | baseline
  duration of professional gaming, daily computer use, game branch, place of competition, and game type
Physical activity status | baseline
  will be classified as active if they engage in ≥150 min/week

CONTACTS AND LOCATIONS:
Locations (1):
- Melike Sumeyye Ozen, Bandırma, Balıkesir, Turkey (Türkiye)